CLINICAL TRIAL: NCT05161364
Title: Analysis of Gait Kinetics in Patients With Foot Dysfunction Either Physiological or Anatomical
Brief Title: Kinetic Analysis Due to Foot Dysfunction
Status: Completed | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Omar Mohamed Ali Elabd, Assistant lecturer, Delta University for Science and Technology
Other Study IDs: 0224786
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2021-12

CONDITIONS: Amputation; Neuropathy;Peripheral
MeSH Terms: conditions — Neuritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: PFA: partial foot amputation secondary to peripheral neuropathy
- B: PN: peripheral neuropathy

SUMMARY:
The aim of the current study is to examine the biomechanical changes of gait kinetics in patients with either partial foot amputation or peripheral neuropathy

ELIGIBILITY:
Inclusion Criteria:

* Partial foot amputees who didn"t receive physiotherapy and don"t use prosthesis. patients with PN grade (1-2) Age 40-65y Both sexes. Walking independently however, no walking aids were used during the testing procedures

Exclusion Criteria:

* Foot amputation levels more proximal than tarso metatarsal joint. Less than 4 months after partial foot amputation. Foot amputees who use prosthesis or suffer from phantom pain. Active foot problems; ulcer, infection, or gangrene. Patients with PN who received physiotherapy or injections like Puerarin Major surgeries in lower limb that could affect either gait or balance like ACL, hip/knee arthroplasty Spine problems that could affect either gait or balance History of ankle sprain. Pathologies such as skin diseases, inflammatory diseases, congenital diseases, or neurological diseases rather than PN.

Fractures or dislocations. Symptomatic degenerative changes that require medications. BMI over 35. Inability of walking independently

Ages: 40 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Convenient 70 patients with 35 patients in each group of both genders ranging in age from 40 to 65 years will participate in this study after examination to exclude any defined pathological conditions. Participants will be recruited from foot amputation centers and outpatient clinics in Mansoura and Damietta, Egypt. All the participants were capable of walking independently to perform their activities of daily life with or without a walking aid. However, no walking aids were used during the testing procedures.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
GRF | 5 minutes
  Ground Reaction Force
Planter Pressure | 3 minutes
  Peak Planter Pressure
Planter Pressure distribution | 4 minutes
  Planter Pressure distribution
Foot surface area | 6 minutes
  Foot surface area

CONTACTS AND LOCATIONS:
Locations (1):
- Delta university, Gamasa, Eldakahlyia, Egypt